CLINICAL TRIAL: NCT01564719
Title: A Randomized Multiple Baseline Intervention Study of Metabolic Syndrome, Mental Health, and Spiritual Well-Being of United Methodist Clergy in North Carolina
Brief Title: Study of a Holistic Health Program for United Methodist Clergy
Acronym: SpiritedLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke Clergy Health Initiative (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Principal Investigator, Rae Jean Proeschold-Bell, Associate Research Professor, Duke University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ORC-1447SP
Record Dates: First submitted 2012-03-14; First posted 2012-03-28 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Depression; Diabetes; Hypertension; Hypercholesterolemia
Keywords: clergy; weight loss; holistic; stress; spiritual
MeSH Terms: conditions — Obesity; Depression; Diabetes Mellitus; Hypertension; Hypercholesterolemia; Weight Loss | interventions — Holistic Health

STUDY DESIGN:
Intervention Model Description: The investigators used a randomized, multiple baseline design in which 3 cohorts were randomly assigned to start date, thereby creating 2 waiting cohorts. Cohort 1 immediately received the intervention; Cohort 2 waited one year and then received the intervention. Cohort 3 waited two years and then received the intervention. Data were collected from Cohorts 2 and 3 while waiting.
Who Masked: Outcomes Assessor
Masking Description: Assessors of metabolic syndrome indicators did not know participants' treatment group.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immediate-intervention arm (Experimental): This is a holistic health intervention. The stress reduction program Williams LifeSkills, adapted for clergy; the 10-session online weight loss program Naturally Slim Foundations plus its 7-session online booster program, Naturally Slim Advanced; monthly phone conversations with Wellness Advocates who function as health coaches; and three in-person workshops that cover the theology of the body and incarnation and provide the religious rationale for caring for the mind and body.
  Interventions: Behavioral: Holistic health
- One-year waitlist arm (Experimental): This holistic health intervention arm for Cohort 2 was the same as Cohort 1's, only the intervention delivery was smoother (e.g., Naturally Slim offered at more start times). Cohort 2 waited for one year before beginning the intervention.
  Interventions: Behavioral: Holistic health
- Two-year waitlist arm (Experimental): This holistic health intervention arm for Cohort 3 was the same as Cohort 2's, only Cohort 3 waited for two years and received the stress management program meQuilibrium rather than Williams LifeSkills.
  Interventions: Behavioral: Holistic health

INTERVENTIONS:
Behavioral: Holistic health — The investigators conceptualize this as a holistic health intervention because it has components involving the mind, body, and spirit. The stress reduction program Williams LifeSkills, adapted for clergy; the 10-session online weight loss program Naturally Slim Foundations plus its 7-session online booster program, Naturally Slim Advanced; monthly phone conversations with Wellness Advocates who function as health coaches; $500 small grants to use to promote health; and three in-person workshops that cover the theology of the body and incarnation and provide the religious rationale for caring for the mind and body.
  Other Names: Williams Life Skills; Naturally Slim

SUMMARY:
This study seeks to test a two-year intervention designed for United Methodist clergy. The intervention consists of: the stress reduction program Williams LifeSkills, adapted for clergy; the 10-session online weight loss program Naturally Slim Foundations plus its 7-session online booster program, Naturally Slim Advanced; monthly phone conversations with Wellness Advocates who function as health coaches; and three in-person workshops that cover the theology of the body and incarnation and provide the religious rationale for caring for the mind and body. Participants were randomly assigned to one of three cohorts, all of which will eventually receive the intervention but which differ by intervention timing, thereby building in a randomized waitlist control group. The investigators hypothesize that intervention participants will achieve reductions in metabolic syndrome, depression, and stress, and achieve improvements in quality of life and spiritual well-being, compared to the waiting control group participants.

DETAILED DESCRIPTION:
Studies are beginning to surface that indicate that clergy suffer from high rates of chronic disease, including obesity (1, 2) and diabetes, arthritis, and hypertension (1). Clergy also experience above average rates of depression (3-5) and anxiety (3, 6). High stress is an additional common problem for clergy. A review of the literature on clergy stress cites the following five stressors as the most salient for clergy: mobility, low financial compensation, inadequate social support, high time demands, and intrusions on family boundaries (7). Health interventions for clergy are needed, and yet, as far as the investigators know, no clergy health interventions have been rigorously tested.

The investigators seek to design and rigorously test a holistic health intervention for United Methodist clergy in North Carolina. Based on the existing epidemiological data, the investigators hope to create a health intervention that will reduce Metabolic Syndrome, which is a set of risk factors that clusters with obesity and is related to cardiovascular disease, diabetes, and death (8, 9). Thus, the investigators seek to reduce rates of hypertension, diabetes, large abdominal circumference, high triglycerides, and low HDL. The investigators additionally seek to decrease stress, depression, and anxiety in clergy.

The investigators developed a 23-month intervention called Spirited Life. This intervention utilizes a combination of: 1) in-person workshops, 2) online videos, 3) contacts with a Wellness Advocate, and 4) small grants. 1) The workshops include the stress management program called Williams LifeSkills, which has a strong evidence base [see, for example, (10)]. The workshops also emphasize theological reasons to take care of one's health. 2) The online videos are the Naturally Slim weight loss and healthy eating program offered by ACAP Health. 3) The Wellness Advocates use Motivational Interviewing to work with clergy to set goals and check on progress. The frequency of Wellness Advocate contact may vary but is intended to be monthly, and generally occurs by phone. 4) The small grants are $500 offered during month 13 of the program and may be broadly used to promote health; participants submit a short application that must be approved by their Wellness Advocate.

The investigators will recruit clergy (Elders, Probationary Elders, Deacons, Interim Supply Pastors, and Local Pastors) serving a local church, as Bishop or as a District Superintendent, or as a campus minister or someone on Conference staff, in either the North Carolina Annual Conference or Western North Carolina Conference, as of July 2010. Additional inclusion criteria are that clergy must be age 18 or higher, and may be full or part-time pastors; student pastors; of any current health status; and non-United Methodist if they are serving a United Methodist Church in one of the North Carolina Conferences. The investigators will exclude extension ministers other than Conference staff and campus ministers, and the investigators will exclude pastors on leave.

This study employs a randomized multiple baseline research design in which all consenting clergy will be randomized to one of three cohorts, which differ in when they will begin receiving the 23-month intervention treatment. Cohort 1 will begin the intervention in January 2011; Cohort 2 in January 2012; and Cohort 3 in January 2013. As is standard in Multiple Baseline research designs, participants in all cohorts will participate in data collection throughout the study period, including prior to their initiation of the intervention treatment.

The investigators will collect both survey and health screening data. The survey data cover the following constructs: depression, anxiety, stress, life satisfaction, relationship satisfaction, hostility, mental and physical health functioning, burnout, spiritual well-being, nutrition, and exercise. The health screening data include height, weight, abdominal circumference, resting blood pressure and heart rate, fasting cholesterol, and hemoglobin A1c.

The data collection schedule varies by cohort, and both survey and health screening data will be sought at each data collection time point. All cohorts will provide baseline survey and health screening data in November 2010. During the 23-month intervention treatment period for each cohort, the investigators will seek data in months 9, 16, and 23. For Cohort 1, the investigators will also seek post-treatment data 6, 12, and 18 months after the end of the intervention period to examine the durability of effects. The investigators will do the same for Cohorts 2 and 3, dependent upon funding.

The investigators' primary analysis will be to compare Cohort 1 at the end of treatment to Cohort 3, which will provide data while waiting for treatment. Thus, embedded in this randomized multiple baseline design is a randomized controlled trial between Cohorts 1 and 3. The investigators therefore will seek data from Cohorts 1 and 3 in September 2011, April 2012, and November 2012. The investigators will also seek data from Cohort 2 in November 2011 to get updated baseline data before Cohort 2 participants start the intervention treatment.

If successful in reducing Metabolic Syndrome, stress, depression, and anxiety, the Spirited Life intervention could have a major impact in reducing health problems and improving the holistic health of clergy.

ELIGIBILITY:
Inclusion Criteria:

* United Methodist Church pastors (Elders, Probationary Elders, Deacons, Interim Supply Pastors, and Local Pastors) serving a local church, as Bishop, as a District Superintendent, or on Conference staff, in either the North Carolina Annual Conference or Western North Carolina Conference as of July 2010
* age 18 or above

Exclusion Criteria:

* Extension ministers other than Conference staff
* Pastors on leave

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Metabolic Syndrome | 2.0 years, 2.5 years, 3.0 years, and 3.5 years
  Changes in abdominal circumference, blood pressure, HbA1c, triglycerides, and HDL. Metabolic Syndrome is defined as having a large abdominal circumference plus two of more of these indicators. We seek to improve each of the five indicators and decrease overall rates of Metabolic Syndrome.

SECONDARY OUTCOMES:
Depression | 2.0 years, 2.5 years, 3.0 years, 3.5 years
  Changes in depression scores measured by the Patient Health Questionnaire-9
Stress | 2.0 years, 2.5 years, 3.0 years, 3.5 years
  Changes in stress scores using the Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: David Toole, PhD, MTS, Principal Investigator — Duke Divinity School; Rae Jean Proeschold-Bell, PhD, Study Director — Duke University
Locations (1):
- Duke Divinity School, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proeschold-Bell RJ, LeGrand SH. High rates of obesity and chronic disease among United Methodist clergy. Obesity (Silver Spring). 2010 Sep;18(9):1867-70. doi: 10.1038/oby.2010.102. Epub 2010 May 6. PMID 20448538
- [Background] Proeschold-Bell RJ, Legrand S, James J, Wallace A, Adams C, Toole D. A theoretical model of the holistic health of United Methodist clergy. J Relig Health. 2011 Sep;50(3):700-20. doi: 10.1007/s10943-009-9250-1. Epub 2009 Apr 10. PMID 19360471
- [Background] Mottillo S, Filion KB, Genest J, Joseph L, Pilote L, Poirier P, Rinfret S, Schiffrin EL, Eisenberg MJ. The metabolic syndrome and cardiovascular risk a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Sep 28;56(14):1113-32. doi: 10.1016/j.jacc.2010.05.034. PMID 20863953
- [Background] Alberti KG, Zimmet P, Shaw J. Metabolic syndrome--a new world-wide definition. A Consensus Statement from the International Diabetes Federation. Diabet Med. 2006 May;23(5):469-80. doi: 10.1111/j.1464-5491.2006.01858.x. PMID 16681555
- [Background] Kirby ED, Williams VP, Hocking MC, Lane JD, Williams RB. Psychosocial benefits of three formats of a standardized behavioral stress management program. Psychosom Med. 2006 Nov-Dec;68(6):816-23. doi: 10.1097/01.psy.0000238452.81926.d3. PMID 17132834
- [Background] Morris ML, Blanton PW. The influence of work-related stressors on clergy husbands and their wives. Family Relations. 1994;43(2):189-95.
- [Background] Jones SH, Francis LJ, Jackson C. The relationship between religion and anxiety: a study among Anglican clergymen and clergywomen. Journal of Psychology & Theology. 2004;32(2):137-42.
- [Background] Halaas GW. Ministerial health and wellness, 2002, Evangelical Lutheran Church in America. Chicago, IL; 2002.
- [Background] Knox S, Virginia SG, Lombardo J. Depression and anxiety in Roman Catholic secular clergy. Pastoral Psychology. 2002;50:345-58.
- [Background] Knox S, Virginia SG, Smith J. Pilot study of psychopathology among Roman Catholic secular clergy. Pastoral Psychology. 2007;55(297-306).
- [Background] Knox S, Virginia SG, Thull J, Lombardo JP. Depression and contributors to vocational satisfaction in Roman Catholic secular clergy. Pastoral Psychology. 2005;54(139-153).
- [Derived] Proeschold-Bell RJ, Turner EL, Bennett GG, Yao J, Li XF, Eagle DE, Meyer RA, Williams RB, Swift RY, Moore HE, Kolkin MA, Weisner CC, Rugani KM, Hough HJ, Williams VP, Toole DC. A 2-Year Holistic Health and Stress Intervention: Results of an RCT in Clergy. Am J Prev Med. 2017 Sep;53(3):290-299. doi: 10.1016/j.amepre.2017.04.009. Epub 2017 Jun 19. PMID 28641912